CLINICAL TRIAL: NCT00372437
Title: A Phase I/II Study of MGCD0103 (MG-0103) in Combination With Gemcitabine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0103-006
Record Dates: First submitted 2006-09-05; First posted 2006-09-07 (Estimated); Last update posted 2015-07-01 (Estimated); Status verified 2015-06

CONDITIONS: Tumors
Keywords: Refractory solid tumors; Phase I/II; Refractory and solid tumors
MeSH Terms: conditions — Neoplasms | interventions — mocetinostat; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: MGCD0103; Drug: Gemcitabine

INTERVENTIONS:
Drug: MGCD0103 — MGCD0103 as an oral dose three times per week.
Drug: Gemcitabine — Gemcitabine 1000mg/m<2> intravenously days 1, 8, 15 of a 28 day cycle.

SUMMARY:
Inthis study, MGCD0103, a new anticancer drug under investigation, is given three times weekly in combination with gemcitabine to patients with solid tumours.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented cancer: Phase I--solid tumors where gemcitabine is considered standard of care; refractory solid tumor with no reasonable likelihood of achieving clinical benefit with existing therapies, that has failed to respond to standard therapy, has progressed despite standard therapy, or for which no standard therapy exists. Phase II--locally advanced and measurable (non-resectable III) or metastatic (Stage IV) pancreatic cancer.
* Patients with known CNS metastases may be enrolled on Phase I or II only if they meet the following criteria:

  * They have received radiotherapy for their CNS disease;
  * They have had steroids discontinued for at least 1 month prior to study entry;
  * They have had a CT or MRI of the brain within 1 month of study entry that shows stable disease; and d)they are free of neurological symptoms.
* Karnofsky performance status of 70 or greater.
* Age 18 years and over.
* Laboratory requirements (must be done within 14 days prior to study initiation):

  * Hematology: White Blood Cells (WBC)≥3 x 10<9>/L (≥ 3000/mm3);
  * Absolute Neutrophil Count (ANC) ≥1.5 x 10<9>/L (≥1500/mm3);
  * Platelets ≥100 x 10<9>/L (≥100,000/mm3);
  * Chemistry: Total Bilirubin ≤1.5 x Upper Limit of Normal(ULN);
  * AST(SGOT)and ALT(SGPT)≤3 x ULN; ≤ 5 x ULN if documented liver metastases;
  * Serum Creatinine ≤1.5 x ULN or calculated creatinine clearance ≥50 mL/min;
  * Urinalysis: Proteinuria <1 mg/dl or 500 mg protein/24 hours if dipstick ≥2+.
* Patients or their legal representative must be able to read (or have read to them), understand, and sign a written informed consent (approved by the institutional review board/Ethics Committee (IRB/EC)) within 14 days prior to start of treatment.

Exclusion Criteria:

* Patients with another active cancer (excluding basal cell carcinoma or cervical intraepithelial neoplasia (CIN/cervical in situ or melanoma in situ). (Phase II portion only)
* Pregnant or lactating women. Women of child bearing potential (WOCBP) must have a negative serum pregnancy test documented within 7 days prior to starting study drug.
* WOCBP and men whose partners are WOCBP must use an acceptable method of contraception while enrolled on this study, and for a period of 3 months following study drug treatment. Patients unwilling or unable to follow this guideline will be excluded. Investigators should follow their Institutional standard regarding acceptable methods of contraception.
* Patients with uncontrolled concomitant illness, active infection requiring i.v. antibiotics, or uncontrolled infections, or a fever >38.5C on the day of scheduled dosing.
* Patients with serious illnesses, medical conditions, or other medical history, including laboratory results, which, in the investigator's opinion, would be likely to interfere with a patient's participation in the study, or with the interpretation of the results.
* Patients who have been treated with any investigational drug within 28 days prior to study initiation (an investigational drug is one for which there is no approved indication), or who are receiving concurrent treatment with other experimental drugs or anti-cancer therapy.
* Known hypersensitivity to HDAC inhibitors or to any of the components of MG-0103.
* Known hypersensitivity to gemcitabine.
* Prior treatment with gemcitabine (during the expanded phase II portion only).
* Known HIV or known active Hepatitis B or C.
* Any condition (e.g., known or suspected poor compliance, psychological instability, geographical location, etc.) that, in the judgment of the investigator, may affect the patient's ability to sign the informed consent and undergo study procedures.
* Any condition that will put the patient at undue risk or discomfort as a result of adherence to study procedures. For example, consider requirement to take MG-0103 with a low pH drink and recommendation to avoid agents that increase gastric pH.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose in combination with azacitidine | 1 year (anticipated)
Response rate | 1 year (anticipated)

SECONDARY OUTCOMES:
Objective response. | 1 year (anticipated)
Pharmacodynamics (histone acetylation, biomarkers) | 1 year (anticipated)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Reid, MSc, MBA, Study Director — MethylGene Inc.
Locations (8):
- United States (6):
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Veterans Affairs Medical Center, Kansas City, Kansas
  - Duke University Medical Center, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Pennsylvania Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
- Canada (2):
  - McGill University/Dept Oncology, Montreal, Quebec
  - CHUS Hopital Fleurimont, Sherbrooke, Quebec